CLINICAL TRIAL: NCT00911144
Title: Booster Vaccination With Pneumococcal Vaccine GSK1024850A or Prevenar™ Co-administered With Hiberix™ in Children Primed With the Same Vaccines
Brief Title: Booster Vaccination Study With a Pneumococcal Vaccine in Children Primed With the Same Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 112933
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Results first posted 2011-01-19 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2016-10

CONDITIONS: Infections, Streptococcal
Keywords: Safety; Pneumococcal vaccine; Immunogenicity; Pneumococcal disease; Booster vaccination
MeSH Terms: conditions — Streptococcal Infections; Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Synflorix Group (Experimental): Subjects previously primed (NCT00680914) with 3 doses of Synflorix and Hiberix in the first year of life receiving a booster dose of the same vaccines in the second year of life by intramuscular injection into the right and the left thigh or deltoid, respectively.
  Interventions: Biological: GSK Biologicals' Synflorix™ (Pneumococcal vaccine GSK1024850A); Biological: GSK Biologicals' Hiberix™
- Prevenar Group (Active Comparator): Subjects previously primed (NCT00680914) with 3 doses of Prevenar and Hiberix in the first year of life receiving a booster dose of Prevenar and Hiberix in the second year of life by intramuscular injection into the right and the left thigh or deltoid, respectively.
  Interventions: Biological: Wyeth-Lederle's Prevenar™; Biological: GSK Biologicals' Hiberix™

INTERVENTIONS:
Biological: GSK Biologicals' Synflorix™ (Pneumococcal vaccine GSK1024850A) — Intramuscular injection, administered as a single dose
  Other Names: Pneumococcal vaccine GSK1024850A
  Arms: Synflorix Group
Biological: Wyeth-Lederle's Prevenar™ — Intramuscular injection, administered as a single dose
  Arms: Prevenar Group
Biological: GSK Biologicals' Hiberix™ — Intramuscular injection, administered as a single dose
  Other Names: Hib

SUMMARY:
The purpose of this study is to evaluate the reactogenicity, safety and immunogenicity of a booster (fourth) dose of pneumococcal vaccine GSK1024850A when co-administered with Hiberix at 12-18 months of age, in children primed with the same vaccines in primary study NCT00680914.

ELIGIBILITY:
Inclusion Criteria:

* A male or female between, and including, 12-18 months of age at the time of booster vaccination.
* Subjects for whom the investigator believes that their parent(s)/ guardian(s) can and will comply with the requirements of the protocol.
* Subjects who received three doses of pneumococcal conjugate vaccine in study NCT00680914.
* Written informed consent obtained from the parent(s)/guardian(s) of the child/ward.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding the vaccination, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to vaccination.
* Administration of immunoglobulins and/or any blood products within three months preceding the vaccination or planned administration during the study period.
* Administration of any pneumococcal and/or Hib vaccine since the end of study NCT00680914.
* Planned administration/administration of a vaccine not allowed by the study protocol during the period starting 1 month (30 days) before the administration of the booster dose of the study vaccines (Visit 1) and up to the follow-up visit (Visit 2) with the exception of vaccines included in the Korean routine immunization which can be given at least one week before the administration of the study vaccines or after study end.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of reactions or allergic disease likely to be exacerbated by any component of the study vaccines.
* Known hypersensitivity to any component of the study vaccines including anaphylactic reactions following the administration of the study vaccines.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Tympanic or axillary/ oral temperature >= 37.5°C or rectal temperature >= 38.0°C. A temperature greater than or equal to these cut-offs warrants deferral of the vaccination pending recovery of the subject.
* Acute disease at the time of enrolment.

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 450 (Actual)
Dates: Start 2009-06-11; Primary Completion 2010-01-11 (Actual); Study Completion 2010-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- South Korea (12):
  - GSK Investigational Site, Ansan
  - GSK Investigational Site, Bucheon-Si, GyeongGi-do,
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, GyeongSangNam-do
  - GSK Investigational Site, Iksan
  - GSK Investigational Site, Jeju City
  - GSK Investigational Site, Jeonju Jeonbuk
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon City, Gyeonggi-do
  - GSK Investigational Site, Wonju-si Kangwon-do

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Kim CH, Kim JS, Cha SH, Kim KN, Kim JD, Lee KY, Kim HM, Kim JH, Hyuk S, Hong JY, Park SE, Kim YK, Kim NH, Fanic A, Borys D, Ruiz-Guinazu J, Moreira M, Schuerman L, Kim KH. Response to primary and booster vaccination with 10-valent pneumococcal nontypeable Haemophilus influenzae protein D conjugate vaccine in Korean infants. Pediatr Infect Dis J. 2011 Dec;30(12):e235-43. doi: 10.1097/INF.0b013e31822a8541. PMID 21817957
- [Background] Kim CH et al. Immunogenicity and safety of 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) in Korean children. Abstract presented at the Korean Society of Pediatric Infectious Diseases - 2011 Spring Conference. Seoul, South Korea, 7-11 June 2011.
- [Background] Kim JS et al. Safety and reactogenicity of booster vaccination with 10-valent pneumococcal non-typeable Haemophilus influenzae protein d conjugate vaccine (PHiD-CV) in Korean children. Abstract presented at the 8th International Symposium on Antimicrobial Agents and Resistance (ISAAR). Seoul, Republic of Korea, 6-8 April 2011.
- [Background] Kim KH et al. Immunogenicity of booster vaccination with 10-valent pneumococcal non-typeable Haemophilus influenzae protein d conjugate vaccine (PHiD-CV) in Korean children. Abstract presented at the 8th International Symposium on Antimicrobial Agents and Resistance (ISAAR). Seoul, Republic of Korea, 6-8 April 2011.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 112933 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112933 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112933 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112933 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112933 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112933 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112933 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two subjects enrolled in the protocol received commercial Prevenar and Hiberix vaccines instead of the clinical vaccines planned to be injected and are as such not included in the number of started subjects below.
Period: Overall Study
Arm/Group | Synflorix Group | Prevenar Group
Started | 335 | 113
Completed | 319 | 108
Not Completed | 16 | 5
Not completed — Withdrawal by Subject | 16 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synflorix Group | Prevenar Group | Total
Number analyzed (Participants) | 335 | 113 | 448
Age, Continuous [Mean (Standard Deviation); unit: months] | 13.6 (1.07) | 13.7 (1.00) | 13.6 (1.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 59 | 227
  Male | 167 | 54 | 221

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Grade 3 Adverse Events
Description: Grade 3 adverse events are severe symptoms that prevent normal, everyday activities.
Time Frame: Within 31 days (Day 0 - Day 30) after booster vaccination.
Population: Analysis was performed on the Total vaccinated cohort on the subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Group | Prevenar Group
Number analyzed (Participants) | 332 | 113
Participants | 42 | 13

2. Secondary Outcome: Number of Subjects Reporting Solicited Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling at the injection site. Solicited general symptoms assessed include drowsiness, fever (equal to or above 37.5 degrees Celsius), irritability and loss of appetite.
Time Frame: Within 4 days (Days 0 to 3) after booster vaccination
Population: Analysis was performed on the Total vaccinated cohort on the subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Group | Prevenar Group
Number analyzed (Participants) | 332 | 113
Participants
  Pain | 120 | 39
  Redness | 142 | 55
  Swelling | 97 | 35
  Drowsiness | 75 | 21
  Fever | 46 | 20
  Irritability | 141 | 42
  Loss of appetite | 71 | 29

3. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events
Description: An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study. Also any "solicited" symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited adverse event.
Time Frame: Within 31 days (Days 0 to 30) after booster vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Group | Prevenar Group
Number analyzed (Participants) | 335 | 113
Participants | 118 | 41

4. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events
Description: Serious adverse events are medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: After booster vaccination up to study end (Month 0 to Month 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Group | Prevenar Group
Number analyzed (Participants) | 335 | 113
Participants | 8 | 4

5. Secondary Outcome: Concentration of Antibodies Against Vaccine Pneumococcal Serotypes
Description: Concentrations of antibodies are measured by 22F-inhibition enzyme-linked immunosorbent assay (ELISA) and are presented as geometric mean concentrations expressed as microgram per milliliter (ug/mL).
  Vaccine pneumococcal serotypes included serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F.
Time Frame: One month after booster vaccination (Month 1)
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data were available for antibodies against at least one study vaccine antigen after booster vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Synflorix Group | Prevenar Group
Number analyzed (Participants) | 317 | 102
ug/mL
  Anti-1: number analyzed (Participants) | 317 | 100
  Anti-1 | 4.03 [3.66 to 4.43] | 0.06 [0.05 to 0.07]
  Anti-4 | 5.77 [5.25 to 6.34] | 12.19 [10.11 to 14.69]
  Anti-5 | 5.51 [5.08 to 5.98] | 0.19 [0.16 to 0.23]
  Anti-6B | 2.78 [2.48 to 3.12] | 7.09 [5.82 to 8.63]
  Anti-7F | 5.39 [4.97 to 5.85] | 0.06 [0.04 to 0.07]
  Anti-9V | 4.99 [4.55 to 5.46] | 12.72 [10.86 to 14.88]
  Anti-14 | 7.73 [7.09 to 8.43] | 22.22 [18.96 to 26.03]
  Anti-18C | 13.14 [11.90 to 14.52] | 14.53 [12.10 to 17.44]
  Anti-19F: number analyzed (Participants) | 317 | 101
  Anti-19F | 16.89 [14.87 to 19.20] | 4.82 [3.97 to 5.85]
  Anti-23F | 3.75 [3.37 to 4.16] | 14.81 [11.61 to 18.89]

6. Secondary Outcome: Opsonophagocytic Activity Against Vaccine Pneumococcal Serotypes
Description: Streptococcus pneumoniae opsonophagocytic activity was measured by a killing-assay using a HL 60 cell line. The results are presented as the dilution of serum (opsonic titer) able to sustain 50% killing of live pneumococci under the assay conditions.
  Vaccine pneumococcal serotypes included serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F.
Time Frame: One month after booster vaccination (Month 1)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Synflorix Group | Prevenar Group
Number analyzed (Participants) | 151 | 47
titer
  Opsono-1: number analyzed (Participants) | 148 | 47
  Opsono-1 | 363.7 [275.3 to 480.5] | 4.7 [3.9 to 5.6]
  Opsono-4: number analyzed (Participants) | 149 | 45
  Opsono-4 | 1058.0 [893.9 to 1252.3] | 3717.0 [2759.3 to 5007.0]
  Opsono-5: number analyzed (Participants) | 150 | 46
  Opsono-5 | 233.9 [189.8 to 288.3] | 4.0 [4.0 to 4.0]
  Opsono-6B: number analyzed (Participants) | 150 | 46
  Opsono-6B | 546.5 [415.9 to 718.0] | 3826.8 [2518.0 to 5815.9]
  Opsono-7F: number analyzed (Participants) | 145 | 46
  Opsono-7F | 5467.5 [4698.1 to 6363.0] | 1038.2 [609.9 to 1767.2]
  Opsono-9V: number analyzed (Participants) | 151 | 44
  Opsono-9V | 1707.5 [1497.6 to 1946.8] | 5204.0 [3842.8 to 7047.4]
  Opsono-14: number analyzed (Participants) | 150 | 46
  Opsono-14 | 1814.6 [1577.4 to 2087.5] | 3958.4 [2888.1 to 5425.4]
  Opsono-18C: number analyzed (Participants) | 147 | 45
  Opsono-18C | 607.9 [498.2 to 741.6] | 1723.3 [1196.4 to 2482.3]
  Opsono-19F: number analyzed (Participants) | 149 | 44
  Opsono-19F | 1284.5 [1027.2 to 1606.3] | 277.3 [171.6 to 448.2]
  Opsono-23F: number analyzed (Participants) | 149 | 44
  Opsono-23F | 2702.9 [2234.9 to 3268.9] | 29918.6 [17115.7 to 52298.1]

7. Secondary Outcome: Concentration of Antibodies Against Cross-reactive Pneumococcal Serotypes 6A and 19A
Description: Concentrations of antibodies are measured by 22F-inhibition ELISA and are presented as geometric mean concentrations expressed as microgram per milliliter.
Time Frame: One month after booster vaccination (Month 1)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Synflorix Group | Prevenar Group
Number analyzed (Participants) | 317 | 102
ug/mL
  Anti-6A | 0.99 [0.84 to 1.17] | 2.51 [1.79 to 3.51]
  Anti-19A | 1.54 [1.27 to 1.87] | 0.32 [0.24 to 0.43]

8. Secondary Outcome: Opsonophagocytic Activity Against Cross-reactive Pneumococcal Serotypes 6A and 19A
Description: Streptococcus pneumoniae opsonophagocytic activity was measured by a killing-assay using a HL 60 cell line. The results are presented as the dilution of serum (opsonic titer) able to sustain 50% killing of live pneumococci under the assay conditions.
Time Frame: One month after booster vaccination (Month 1)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Synflorix Group | Prevenar Group
Number analyzed (Participants) | 146 | 44
titer
  Opsono-6A: number analyzed (Participants) | 137 | 44
  Opsono-6A | 196.1 [134.6 to 285.9] | 1415.7 [891.2 to 2248.9]
  Opsono-19A | 64.9 [44.6 to 94.5] | 15.5 [8.1 to 29.9]

9. Secondary Outcome: Concentration of Antibodies Against Protein D (PD)
Description: Concentrations of antibodies are presented as geometric mean concentrations expressed as Enzyme-Linked Immuno-Sorbent Assay (ELISA) units per milliliter (EU/mL).
Time Frame: One month after booster vaccination (Month 1)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Synflorix Group | Prevenar Group
Number analyzed (Participants) | 316 | 101
EU/mL | 1288.9 [1175.6 to 1413.2] | 92.0 [78.3 to 108.1]

10. Secondary Outcome: Concentration of Antibodies Against Polyribosyl-ribitol-phosphate (PRP)
Description: Concentrations of antibodies are presented as geometric mean concentrations expressed as microgram per milliliter.
Time Frame: One month after booster vaccination (Month 1)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Synflorix Group | Prevenar Group
Number analyzed (Participants) | 163 | 54
ug/mL | 152.970 [130.307 to 179.575] | 99.738 [72.964 to 136.335]

ADVERSE EVENTS:
Time Frame: Serious AEs were assessed up to one month following booster vaccination (Month 1). The time frames for Other AEs reporting were 4 days and 31 days following booster vaccination for events collected by systematic and non-systematic methods, respectively.
Description: Subjects at risk for systematically assessed other (non-serious) adverse events has been set to the number of subjects that had returned their symptom sheet.
Arm/Group | Synflorix Group | Prevenar Group
Serious Adverse Events (participants affected / at risk) | 8/335 | 4/113
Other Adverse Events (participants affected / at risk) | 243/335 | 82/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix Group (N=335) | Prevenar Group (N=113)
Pharyngitis (Infections and infestations) | 0 | 2
Pharyngotonsillitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 2 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Febrile convulsion (Nervous system disorders) | 1 | 0
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0
H1N1 influenza (Infections and infestations) | 1 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 1 | 0
Otitis media acute (Infections and infestations) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Synflorix Group (N=335) | Prevenar Group (N=113)
Upper respiratory tract infection (Infections and infestations) | 30 | 12
Nasopharyngitis (Infections and infestations) | 19 | 10
Pain at the injection site (General disorders) | 120/332 | 39
Redness at the injection site (General disorders) | 142/332 | 55
Swelling at the injection site (General disorders) | 97/332 | 35
Drowsiness (General disorders) | 75/332 | 21
Fever (General disorders) | 46/332 | 20
Irritability (General disorders) | 141/332 | 42
Loss of appetite (General disorders) | 71/332 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.